CLINICAL TRIAL: NCT01744054
Title: Pilot Study of Microsphere Localization Using PET/MRI or PET/CT in Patients Following Radioembolization
Brief Title: Microsphere Localization Using PET/MRI or PET/CT in Patients Following Radioembolization
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Logistics regarding PET/CT portion of study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201209062
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET/MR or PET/CT (Other): * Patients must have had radioembolization, within 72 hours of the PET/MR or PET/CT
  * Subjects will be asked to lie still within the scanner for up to 1.5 hours while images are acquired for the liver
  Interventions: Device: PET/MR; Device: PET/CT

INTERVENTIONS:
Device: PET/MR
Device: PET/CT

SUMMARY:
The successful localization of the y90 microspheres by PET/MR and/or PET/CT scans would be a useful tool in individualizing patient care after the radioembolization procedure. The information from a PET/MR or PET/CT scan would allow for early evaluation of the technical success of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant must successfully complete the MRI screening form if receiving an MRI
* Participant must be scheduled to undergo radioembolization for any indication
* Participant must be ≥ 18 years of age
* Participant must be able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent document

Exclusion Criteria:

* Participant must not have any contraindications to MRI scanning
* Patient must not be pregnant or breastfeeding
* If agreeing to MRI contrast, participant must not have renal insufficiency (glomerular filtration rate (GFR < 30 mL/min/1.73 m2) measured within the past 60 days
* If agreeing to MRI contrast, participant must not be on dialysis
* If agreeing to MRI contrast, participant must not have had a prior allergic reaction to gadolinium-based contrast agents
* PET/MRI or PET/CT is not able to be scheduled within 72 hours of radioembolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10-25 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Evaluate y90-PET/MRI and PET/CT for potential on reporting presence of extrahepatic deposition of microspheres | 1 day (one time event for patient)
  A diagnostic radiologist and a nuclear medicine physician will evaluate the images and will determine any presence of extrahepatic deposition of microspheres.
Evaluate y90-PET/MRI and PET/CT for potential on reporting technical success of radioembolization | 1 day (one time event for patient)
  A diagnostic radiologist and a nuclear medicine physician will evaluate the images and will determine whether technical success of the procedure can be determined. They will rate the images if they are 'adequate' to report on these two measures.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu